## INFORMED FOR BODY BLOCK APPLICATIONS VOLUNTEER CONSENT FORM

Study Title: Comparison of the Effects of TAP (Transversus Abdominis Plan) Block and QLB-1 (Lateral Quadratum Lumbarum) Block on Postoperative Pain and Opioid Consumption in Laparoscopic Cholecystectomy Operations

| Number of Volu | nteers: 60 |
|-------------------|--------------|
| Research Duration | on: 6 months |
| Date | : / / |
| Name-Surname | : |
| Telephone | : |

Body Block application approved.....

You are voluntarily participating in our research on 'Comparison of the superiority of different preoperative trunk blocks for postoperative pain control in closed gallbladder surgery'. Our aim is to find a more effective analgesia method with fewer side effects after closed abdominal surgery. There are two different groups in the study and you will be randomly selected which group you will be included in. Torso blocks are a comfortable analgesia method created by injecting a local anesthetic into the plane of the abdominal muscles with a thin needle under ultrasound guidance so that patients who will undergo abdominal surgery do not feel pain during and especially after surgery. The local anesthetic is injected into a specific muscle plane and is aimed to reach and spread to the nerves. The appropriate abdominal area to be injected and the ultrasound probe will be cleaned with the necessary materials and the ultrasound probe will be placed parallel to the abdomen. The muscles and abdominal cavity will be easily visualized and under germ-free conditions, a thin needle will be inserted through the skin and the appropriate medication will be injected as needed. If you are allergic to any medication, please inform your doctor before the procedure. Although you have not been allergic before, allergic events may still occur during the procedure. All kinds of medicines and equipment are available to treat allergic events during the procedure. However, despite treatment, respiration and blood circulation may stop as a result of a severe allergic reaction and intensive care may be required. Again, the drugs used during the applications may slow down your breathing, heart rate and lower your blood pressure. As a precaution, your blood pressure and heart rate will be monitored with a monitor.

| Patient's Name and Surname: | Date and Signature |
|-------------------------------------------------|--------------------|
| Practicing Doctor: | Date and Signature |
| Specialist Dr. Emine ÖZCAN | |
| Tel: +90 530 159 28 56 (available 24/7) | |
| Name and Surname of the person or institutional | Date and Signature |
| official who witnessed the consent process from | |
| beginning to end: | |

Necessary blood tests will be performed before the procedures. However, the risk of bleeding increases especially in patients who use anticoagulants (blood thinners). The use of blood thinners before the procedure should be discontinued under the control of your doctor. The procedures will be postponed until the bleeding tests are at the appropriate level. Please inform your doctor if you are taking such medications.

## Problems that may arise during or after body blocks:

- **Problems related to block type:** There will be two different types of blocks in the study and you will be randomly assigned which block to do. Since our aim is to find out which type of block is more effective or superior, there may be differences between the two types of blocks. One block may have better or longer lasting pain relief than the other. It may have different effects on the length of hospital stay. You may need additional pain relief despite the block. In such cases, necessary interventions will be made.
- **Allergy to medication:** You may develop an allergy to the local anesthetics given for the block. Medical intervention will be provided if necessary.
- **Intravenous administration of drugs:** Drugs administered during the block due to their close proximity to the vessels may unintentionally pass into the circulatory system. This may cause dizziness, drowsiness, impaired consciousness, epileptic attacks (epileptic seizures). Medical intervention will be provided if necessary.
- **Bleeding/bruising/hematoma:** Due to the puncture of neighboring vessels, blood may leak from the vessel into the tissue and accumulate in this area.
- **Infection at the site of intervention:** As with any injection, infection may develop in these procedures.
- The pain does not go away or increases: Although it is aimed to relieve or reduce your pain after the procedure, this is not guaranteed. Temporary pain at the injection site or an increase in pre-existing pain may be possible after the procedure.
- **Injury to organs on the needle entry and exit route:** There may be injuries to the peritoneum, liver, intestine. However, we do not encounter these with the use of ultrasound.

| Patient's Name and Surname: | Date and Signature |
|---|---|
| Practicing Doctor: Specialist Dr. Emine ÖZCAN Tel: +90 530 159 28 56 (available 24/7) | Date and Signature |
| Name and Surname of the person or institutional official who witnessed the consent process from beginning to end: | Date and Signature |

I have read all possible side effects of the above-mentioned treatment and/or interventions planned to be applied to me, and all explanations in the informed consent form. Written and verbal explanations about the research, the subject and purpose of which are stated above, were made to me by the physician named below. I know that I am participating in the research voluntarily and that I can leave the research at any time with or without justification.

I understand the information given to me, the possibility of ineffective treatment, the possible effects, side effects, complications, risks of the method or medication to be applied, and all medical interventions that may be made by my doctor during the prevention or treatment of these, and I agree to participate in the research in question with my own consent, without any pressure or coercion, under the witness of my relative and the doctor mentioned below.

| Patient's Name and Surname: | Date and Signature |
|---|---|
| Practicing Doctor: Specialist Dr. Emine ÖZCAN Tel: +90 530 159 28 56 (available 24/7) | Date and Signature |
| Name and Surname of the person or institutional official who witnessed the consent process from beginning to end: | Date and Signature |